CLINICAL TRIAL: NCT01508533
Title: Disease Burden Study and Site Preparation for Planning and Implementation of the Phase III Trials for the Oral Rotavirus Vaccine 116E
Brief Title: Epidemiology of Rotavirus Infection in North India Community
Status: Completed | Type: Observational
Sponsor: Society for Applied Studies (Other)
Collaborators: National Institute of Immunology, New Delhi (Unknown); Ministry of Science and Technology, India (Other Government)
Responsible Party: Principal Investigator, NBhandari, Joint Director, Society for Applied Studies
Other Study IDs: SAS/BBIL/07/2008
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Rotavirus Gastroenteritis
Keywords: Disease burden; Rotavirus gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1: Infants enrolled at ≤1 week and followed up weekly till one year of age.
- Cohort 2: Cohort 2: Infants enrolled at 12 months and followed up weekly till they are aged 24 months.

SUMMARY:
This study was designed to support site preparation and to conduct a disease burden study for the planning and implementation of the phase III trials for the oral rotavirus vaccine 116E.

DETAILED DESCRIPTION:
Field workers conducted weekly surveillance in areas allocated to them and identified pregnant women, newborns and infants aged 9 to 12 months. Children who were eligible for participation through criteria for inclusion and exclusion in the trial were enrolled. Two cohorts were recruited, one cohort enrolled within one week of birth and followed up weekly till 1 year of age (cohort 1=100) and the second cohort enrolled at 12 months of age and followed up till 24 months of age (cohort 2=100).

Weekly contact were made by field workers for both the cohorts. At each contact cases of gastroenteritis were identified. All infants with gastroenteritis were assessed by a field worker/clinical coordinator. The child was assessed for presence of dehydration, danger signs. The field worker/clinical coordinator ensured that at least one diarrheal stool specimen was collected for each episode of gastroenteritis. Infants were treated at the study clinic or escorted to one of the identified hospitals, if required.

Caregivers of the enrolled infants were explained the signs and symptoms of suspected intussusception, dehydration and danger signs that require hospital referral and were given the option to seek care from the study clinic or from one of the identified hospitals in the vicinity.

Stool specimens were collected in all diarrheal episodes. In a subset of 30 children who were identified early in a diarrheal episode and who shed rotavirus, multiple stool specimens were collected in order to assess duration of shedding of rotavirus during a natural infection.

The study was also designed to collect information on data essential for planning and implementation of phase III trials pertaining to trial logistics, data collection tools and validity of questions including those in the Vesikari score.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardian consent for participation and are able to understand study procedures
* Healthy infant aged ≤ 1 week - cohort I, children aged 12 months (+14 days)-Cohort 2
* Absence of any illness requiring hospitalization
* No confirmed plans to move in the next 12 months

Exclusion Criteria:

* Participating in any other trial
* Any signs or symptoms of active sepsis, pneumonia, meningitis or any other disease requiring hospitalization
* Known case of immunodeficiency disease, known HIV positive
* Known case of chronic gastrointestinal disease
* Any other conditions which in the judgment of the investigator warrant exclusion(e.g. no exclusion criteria but seems 'ill', investigators suspects neglect)

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study was conducted in Delhi at Govindpuri-Tigri-Dakshinpuri, Tuglakabad and Sangam Vihar.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Disease burden | 1 year
  All episodes of gastroenteritis:
  * rotavirus gastroenteritis
  * rotavirus gastroenteritis by the G and P types
  * severe gastroenteritis
  * severe rotavirus gastroenteritis
  * severity score of all episodes of gastroenteritis
  Rates of hospitalization in the above categories
  Proportion requiring rehydration therapy in all the above categories
Duration of rotavirus shedding | 1 year
  To ascertain the duration of rotavirus shedding after an episode of rotavirus gastroenteritis
Rotavirus genotypes | 1 year
  To identify genotypes of rotavirus
Data collection for planning and implementation of phase III trials | 1 year
  To collect information on data essential for planning and implementation of phase III trials pertaining to trial logistics, data collection tools and validity of questions including those in the Vesikari score.

CONTACTS AND LOCATIONS:
Overall Officials: Nita Bhandari, PhD, Principal Investigator — Society for Applied Studies
Locations (1):
- Society for Applied Studies, New Delhi, National Capital Territory of Delhi, India